CLINICAL TRIAL: NCT07137351
Title: The Biosensor Using the Target Urine Volatile Organic Compounds for Detecting Diabetic Kidney Disease
Brief Title: The Biosensor Using the Target Urine VOCs for Detecting DKD Diabetic Kidney Disease
Acronym: VOCs in DKD
Status: Withdrawn | Type: Observational
Why Stopped: This record was initially withdrawn due to incomplete protocol section. The study was completed and published, and a corrected version will be submitted under a new record
Sponsor: Suranaree University of Technology (Other)
Responsible Party: Principal Investigator, Chatchai Kreepala, MD, Associate Professor Dr. Chatchai Kreepala, M.D., Suranaree University of Technology
Other Study IDs: EC-67-0001
Record Dates: First submitted 2024-06-07; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Urine VOCs From DKD and Nephrotic Syndrome Pateints
Keywords: VOCs; Biosensor; diabetic kidney disease; nephrotic syndrome
MeSH Terms: conditions — Diabetic Nephropathies; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 3: ็Healthy volunteer, DKD pateints, other causes of Nephrotic syndrome
  Interventions: Diagnostic Test: The Biosensor Using the Target Urine Volatile Organic Compounds
- ็Healthy volunteer: ็Healthy volunteer = normal subject or diabetes pateint without proteinuria (< 300 mg/day)
  Interventions: Diagnostic Test: The Biosensor Using the Target Urine Volatile Organic Compounds
- DKD pateints: DKD = diabetic kidney disease with proteinuria (> 1 g/day) with confirmed by pathological results
  Interventions: Diagnostic Test: The Biosensor Using the Target Urine Volatile Organic Compounds
- other causes of Nephrotic syndome: NS = other casues of nephrotic syndrome, pateints must have with proteinuria > 3.5 g/day) with confirmed by pathological results. In addition, They must have no DM in the illness profile.
  Interventions: Diagnostic Test: The Biosensor Using the Target Urine Volatile Organic Compounds

INTERVENTIONS:
Diagnostic Test: The Biosensor Using the Target Urine Volatile Organic Compounds — The authors opted to utilize five distinct commercially available semiconductors (metal oxide sensors) to detect all the targeted VOCs which were manufactured by Figaro company.
  Urine samples from patients were placed in a urine container, which was then placed into the VOCs detection device. The lid was closed, and the system was set to operate in a closed-loop mode at a room temperature of 25 degrees Celsius. The device then vacuumed VOCs from the urine samples of the patients through a gas tube into the biosensor chamber located on top, where analysis was performed.
  Other Names: Metal oxide semiconductor detecting VOCs

SUMMARY:
Volatile organic compounds (VOCs) are easily evaporated substances produced by pathophysiologic metabolism and have been utilized in research as potential new biomarkers for differentiating various diseases, acting as the odor imprints of each disease.

Researchers used metal oxide semiconductors to examine the properties of VOCs produced by diabetic kidney disease patients. Also, the VOCs of those with diabetic kidney disease were then compared with those of healthy individuals and patients with nephrotic syndrome.

The study found that VOCs primarily composed of hydrogen, methanol, and sulfate in diabetic kidney disease patients had a significantly different ability to release free electrons from the metal oxide semiconductors compared to healthy individuals and patients with nephrotic syndrome from other causes. This finding suggested that VOCs could be used as biomarkers which could lead to the replacement of renal biopsy for diagnosis in the future.

DETAILED DESCRIPTION:
This study was a descriptive cohort study. General data such as age, gender, medications, other medical conditions, or chronic diseases that might have affected the urine VOCs test were reviewed and recorded from the medical records of subjects who attended the outpatient clinic of the Internal Medicine department at the Suranaree University of Technology Hospital from March 2024 to July 2024. Urine samples from diabetic patients, both with and without abnormal proteinuria, were compared with normal urine samples and urine samples from patients with NS from other causes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20 years
* In DKD and NS groups must undergone renal biopsy before study

Exclusion Criteria:

* Patients with an estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73 m2
* Pregnancy
* Ambiguous pathological results

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study was a descriptive cohort study. General data such as age, gender, medications, other medical conditions, or chronic diseases that might have affected the urine VOCs test were reviewed and recorded from the medical records of subjects who attended the outpatient clinic of the Internal Medicine department at the Suranaree University of Technology Hospital from March 2024 to July 2024. Urine samples from diabetic patients, both with and without abnormal proteinuria, were compared with normal urine samples and urine samples from patients with NS from other causes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Characteristic of VOCs in DKD | March 2024- July 2024
  Electrical resistance characteristic VOCs by semiconductors in DKD when compared to normal and NS

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medicine, Suranaree University of Technology, Nakhon Ratchasima, Thailand

IPD SHARING:
Plan to Share IPD: No
the urine samples were indentided by some special code and not allowed to share with other researches.